CLINICAL TRIAL: NCT00147004
Title: Corticosteroid Therapy of Septic Shock - Corticus. A Multi-National, Prospective, Double-Blind, Randomized, Placebo-Controlled Study
Brief Title: Corticosteroid Therapy of Septic Shock - Corticus
Acronym: Corticus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: European Society of Intensive Care Medicine (Other); International Sepsis Forum (Other); The Gorham Foundation (Unknown)
Responsible Party: Prof. Charles Sprung, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLK2-CT-2000-00589; EC- QLK2-CT-2000-00589
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Shock, Septic
Keywords: Septic shock; Steroids; Hydrocortisone; Mortality; Reversal of shock; Adrenal insufficiency
MeSH Terms: conditions — Shock, Septic; Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): hydrocortisone sodium succinate
  Interventions: Drug: hydrocortisone sodium succinate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydrocortisone sodium succinate — 50 mg intravenous bolus every six hours for 5 days, then tapered to 50 mg intravenously every 12 hours for days 6-8, 50 mg every 24 hours for days 9-11 and then stopped
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether steroids decrease 28-day mortality in patients with septic shock.

DETAILED DESCRIPTION:
The use of steroids in septic shock remains controversial. The purpose of this study is to determine whether hydrocortisone decreases 28-day mortality in patients with septic shock. The primary end point will be 28-day mortality in all the non-responders to ACTH (< or = 9 mcg/dl or 250 nmol/L post ACTH). Secondary endpoints will be 28 day all cause mortality in the total group and in responders, ICU and hospital mortality, one year mortality, organ system failure reversal especially shock, and duration of ICU and total hospitalisation.

In a double-blinded fashion (randomized on a 1:1 basis), patients receive 50 mg intravenously every 6 hours for 5 days. After 5 days, treatment will be tapered with 50 mg given intravenously every 12 hours for days 6-8, then 50 mg every 24 hours for days 9-11, and then stopped.

All concomitant treatments, including antibiotics, fluids, vasopressors and ancillary therapies will be given at the discretion of the primary care physician. Evidence-based guidelines for the management of severe sepsis and septic shock by the International Sepsis Forum (Intensive Care Med 2001;27:S124-S134) are encouraged to be followed.

All serious adverse events (SAE) which occur between days 0 and 28, which are unexpected and/or considered possibly or probably related to the study medication, must be documented and reported within 24 hours to the Safety and Efficacy Monitoring Committee. Non-serious adverse events will be listed on the case report form if they are unexpected and believed to be related to the study drug during days 0 to 14.

Specific adverse events which will be monitored closely because of their relationship to corticosteroids and shock are:

1. Use of corticosteroids, i.e. gastrointestinal bleeding and superinfection; hyperglycemia, hypernatremia, muscular weakness, etc.
2. Shock and use of vasopressors, i.e. stroke, acute myocardial infarction and peripheral ischemia.

In addition, substudies will include harmonization of cortisol by comparing cortisol levels measured in local laboratories and a central laboratory, immune and neuro-endocrine interactions, neuromuscular weakness and cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical evidence of infection within the previous 72 hours (may be present longer than 72 hours) (a, b, c, or d - only 1 required)

   1. Presence of polymorphonuclear cells in a normally sterile body fluid (excluding blood);
   2. Culture or Gram stain of blood, sputum, urine or normally sterile body fluid positive for a pathogenic micro-organism;
   3. Focus of infection identified by visual inspection (e.g. ruptured bowel with the presence of free air or bowel contents in the abdomen found at the time of surgery, wound with purulent drainage);
   4. Other clinical evidence of infection - treated community acquired pneumonia, purpura fulminans, necrotising fascitis, etc.
2. Evidence of a systemic response to infection as defined by the presence of two or more of the following signs within the previous 24 hours. These signs may be present longer than 72 hours.

   1. Fever (temperature >38.3°C) or hypothermia (rectal temperature < 35.6°C);
   2. Tachycardia (heart rate of >90 beat/min);
   3. Tachypnea (respiratory rate > 20 breaths/min, PaC02<32 mmHg) or patient requires invasive mechanical ventilation;
   4. Alteration of the WBC count >12,000 cells/mm3, <4,000 cells/mm3 or >10% immature neutrophils (bands).
3. Evidence of shock defined by (A + B- both required within the previous 72 hours (may NOT be present longer than 72 hours).

A. A systolic blood pressure < 90 mmHg or a decrease in SBP of more than 50 mmHg from baseline in previous hypertensive patients (for at least one hour) despite adequate fluid replacement OR need for vasopressors for at least one hour (infusion of dopamine ≥ 5 mcg/kg/min or any dose of adrenaline, noradrenaline, phenylephrine or vasopressin) to maintain a SBP ≥ 90 mmHg;

B. Hypoperfusion or organ dysfunction which is not the result of underlying diseases or drugs, but is attributable to sepsis, including one of the following:

1. Sustained oliguria (urine output < 0.5 ml/kg/hr for a minimum of 1 hour)
2. Metabolic acidosis [pH of < 7.3, or a base deficit of > or = 5.0 mmol/L, or an increased lactic acid concentration (> 2 mmol/L)].
3. Arterial hypoxemia (Pa02/FI02<280 in the absence of pneumonia)(Pa02/FI02<200 in the presence of pneumonia).
4. Thrombocytopenia - platelet count ≤ 100,000 cells/mm3.
5. Acute altered mental status (Glasgow Coma Scale < 14 or acute change from baseline).

4. Informed Consent

5. Cortisol level at baseline and 60 minutes after 0.25 mg cosyntropin

Exclusion Criteria:

1. Pregnancy
2. Age less than 18.
3. Underlying disease with a prognosis for survival of less than 3 months.
4. Cardiopulmonary resuscitation within 72 hours before study.
5. Drug-induced immunosuppression, including chemotherapy or radiation therapy within 4 weeks before the study.
6. Administration of chronic corticosteroids in the last 6 months or acute steroid therapy (any dose) within 4 weeks (including inhaled steroids). Topical steroids are not exclusions.
7. HIV positivity.
8. Presence of an advanced directive to withhold or withdraw life sustaining treatment (i.e. DNR).
9. Advanced cancer with a life expectancy less than 3 months.
10. Acute myocardial infarction or pulmonary embolus.
11. Another experimental drug study within the last 30 days.
12. Moribund patients likely to die within 24 hours.
13. Patients in the ICU for more than 2 months at the time of the start of septic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2002-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
28 day mortality in all the non-responders to ACTH (< or = 9 mcg/dl or 250 nmol/L post ACTH) | 28 days

SECONDARY OUTCOMES:
28 day all cause mortality in the total group. | 28 days
28 day all cause mortality in responders. | 28 days
One year mortality in nonresponders, total and responders. | one year
ICU and hospital mortality. | one year
Organ system failure reversal, especially shock. | one year
Duration of ICU and total hospitalisation. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Sprung, MD, Study Chair — Hadasah Medical Organization; Djillali Annane, MD, Study Director — Hopital Raymond Poincare; Josef Briegel, MD, Study Director — Ludwig-Maximilian-Universitaet Muenchen; Didier Keh, MD, Study Director — Charite Campus Virchow-Klinikum; Rui Moreno, MD, Study Director — Hospital de St. António dos Capuchos; Didier Pittet, MD, Study Director — University Hospital, Geneva; Mervyn Singer, MD, Study Director — University College, London
Locations (57):
- Austria (4):
  - LKH Feldkirch, Feldkirch
  - KH-BHS Linz, Linz
  - Krankenhaus der Barmherzigen Schwestern Ges. mbH, Linz
  - Universitaetsklinik fuer Innere Medizin II, Vienna
- Belgium (4):
  - Hopital St. Joseph, Arlon
  - University Hospital Erasme, Brussels
  - Cliniques Universitaires St. Luc, UCL, Brussels
  - CHU Charleroi, Charleroi
- France (6):
  - Hopital Raymond Poincare, Paris, Garches
  - Hopital Lariboisiere, Paris, Oarus
  - Hopital de Caen, Caen
  - Hopital Huriez, Lille
  - Hopital Caremeau, Nîmes
  - Hopital Saint-Antoine, Paris
- Germany (24):
  - Zentralklinikum Augsburg, Augsburg
  - Vivantes-Klinikum im Friedrichshain, Berlin
  - Vivantes-Klinikum Spandau, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Charité Campus Mitte, Berlin
  - St. Joseph Krankenhaus, Berlin
  - Charité - Campus Benjamin Franklin, Berlin
  - Vivantes-Klinikum Neukoelln, Berlin
  - Charité - Campus Charité Mitte, Berlin
  - Charité Campus Virchow -Klinikum, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Charité- Campus Virchow- Klinikum, Berlin
  - Institute for Anaesthesia and Operative Intensive Care, Darmstadt
  - University Hospital Dresden, Dresden
  - Krankenhaus Hennigsdort, Hennigsdorf
  - Friedrich-Schiller Universitaet, Jena
  - Klinikum Kemptern-Oberallegaeu, Kempten
  - Klinikum Landshut, Landshut
  - Klinikum Mannheim, University of Heidelberg, Mannheim
  - Klinikum Grosshadern, LMU Munich, Munich
  - Staedtisches Krankenhaus Muenchen-Harlaching, München
  - Ludwig-Maximilian-Universitaet Muenchen, München
  - Univesitaet Erlangen-Namberg, Nuremberg
  - Klinikum Ernst von Bergman, Potsdam
- Israel (4):
  - Haemek Hospital, Afula
  - Hadassah Medical Organisation, Jerusalem
  - Beilinson Medical Centre, Petah Tikva
  - Ichilov Hospital, Tel Aviv
- Italy (2):
  - Policlinico di Tor Vergata, Roma
  - Centro di Rianimazione Ospedale S.Eugenio, Roma
- Netherlands (2):
  - Renier de Graaf Hospital, Delft
  - Erasmus University Medical Centre, Rotterdam
- Portugal (3):
  - Hospital de St. Antonio do Capuchos, Lisbon
  - UCIP, Hospital de Desterro, Lisbon
  - Hospital de Egas Moniz, Lisbon
- United Kingdom (8):
  - Aberdeen Royal Infirmary, Aberdeen
  - Southend Hospital, Essex
  - Ipswich Hospital, Ipswich
  - Royal Lancaster Infirmary, Lancaster
  - The General Infirmary at Leeds, Leeds
  - Bloomsbury Institute of Intensive Care Medicine, London
  - University of Manchester, Hope Hospital, Salford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Background] Annane D, Briegel J, Sprung CL. Corticosteroid insufficiency in acutely ill patients. N Engl J Med. 2003 May 22;348(21):2157-9. doi: 10.1056/NEJM200305223482123. No abstract available. PMID 12761380
- [Result] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Derived] Polito A, Sonneville R, Guidoux C, Barrett L, Viltart O, Mattot V, Siami S, Lorin de la Grandmaison G, Chretien F, Singer M, Gray F, Annane D, Brouland JP, Sharshar T. Changes in CRH and ACTH synthesis during experimental and human septic shock. PLoS One. 2011;6(11):e25905. doi: 10.1371/journal.pone.0025905. Epub 2011 Nov 3. PMID 22073145